CLINICAL TRIAL: NCT01028118
Title: Domestic and Sexual Violence Against Women: Consequences for Climacteric´s Phase
Brief Title: Violence Against Women and Consequences During Climacteric´s Phase
Acronym: DV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Núcleo de Estudos Sobre Violência e Humanização da Assistencia à Saúde (Other)
Responsible Party: Edmund Chada Baracat, University of Sao Paulo General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 180/09
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2009-03

CONDITIONS: Violence; Battered Women; Cognitive Behavior Therapy
Keywords: domestic and sexual violence; menopause; professional improvement; social support network
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapy for Women reporting violence (Other): Asking about life experience with violence and Cognitive Behavior Therapy.
  Interventions: Other: Identifying experience with violence

INTERVENTIONS:
Other: Identifying experience with violence — Asking about life experience with violence and Cognitive Behavior Therapy.
  Other Names: Violence attention; Therapy

SUMMARY:
Objective- Analysis of the health status of women who were or are victims of domestic and sexual violence seeking attention at the outpatient clinic for Endocrines Gynecology and Climactery - University of Sao Paulo General Hospital.

To widen the comprehension of the binomial relationship violence-pathologies by professionals/staff who work in health services, offering women in such situation humane, comprehensive and qualified attention. Specific Objectives: decreasing the rates of domestic and sexual violence against women employing: prevention, health education and treatment - within the context of health services and public policies.

Methodology - Project Type: Research in Action A- Attention to women in a situation of domestic and sexual violence during climactery; B- Information/Education/Communication (IEC) C- Behavioral Intervention (IC) D- Institutional Development (DI). Target Populations: 1. Women (during the ages of 40 to 65 years) who were or are victims of domestic and/or sexual violence; 2. Professional/staff who work in services attending women in sexual and domestic violent situations (health professionals, policemen, civil society) in areas located within the South Regional Health Coordination - SRC. To collect information, a semi structured questionnaire will be employed during seven months in 2009.

DETAILED DESCRIPTION:
Trained professionals will work in the regions of: Campo Limpo, M'Boi Mirim, Santo Amaro and neighboring regions, neighborhood in which the Social Vulnerability Index of São Paulo (IPVS) shows high records.

ELIGIBILITY:
Inclusion Criteria:

* Women (during the ages of 40 to 65 years) who were or are victims of domestic and/or sexual violence

Exclusion Criteria:

* Women who were not victims of domestic and/or sexual violence.
* Women that were not 40 to 65 years.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Sessions of Cognitive Behavioral Therapy is good for women subject to sexual violence. | 8 months
  Women subjected to sexual violence had significative higher incidence of depression and fibromyalgia that did not respond to classic treatment; after two of Cognitive Behavioral Therapy started to respond to medicine previously employed.
PREVENTION OF DOMESTIC VIOLENCE IN CHILDOOD AND/OR ADOLESCENTS: LESSER PREVALENCE OF COMORBIDITIES IN CLIMACTERIC´S PHASE. | four months
  Analyzing among women who suffered violence in childhood and/or adolescence comorbidities they suffered in climacteric´s phase. We applied a semi-structured questionnaire for women in climactery who suffered domestic violence. We performed descriptive and comparative analysis on violences both groups (violence in childhood and/or adolescence and violence in adulthood) with chronic affections presented in climactery.
  Conclusion: suffering domestic violence during childhood and/or adolescence presents higher prevalence of comorbidities during climacteric´s phase.
Analyzing among women who suffered violence the comorbidities they suffered in climacteric´s phase. | 3 months
  Chronic pathologies in women who suffered violence in childhood/adolescence: Hypertension 47,5%, Diabetes 14,17%, Depression 70,0%;Labyrintitis 36,67%, Fybromialgy 30,83%, Rheumatic disease 25,0%, Ovarian cancer 1,67%, Uterine cancer 3,33%, Disk hernia 13,33%, Allergies 30,83%, Bronchitis 10,83%, Thrombosis 6,67%. Comparing these women to those who suffered violence during adulthood, these women resulted in higher prevalence of Diabetes, Depression, Labyrintitis, Ovarian cancer, Bronchitis/breathing allergies and Thrombosis, when compared to women subjected to violence during adulthood.

SECONDARY OUTCOMES:
Sessions of Cognitive Behavioral Therapy is good for women subject to sexual violence. | 8 months
  Women subjected to violence in any phase of their lives had at least three chronic comorbidities. The correlation between having been subjected to violence and suffering from depression, fibromyalgia or sexual dysfunctions (statistical significant).

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Dircinha TA Moraes, Post-Doc, Principal Investigator — University of Sao Paulo General Hospital; Edmund C Baracat, Titular Prof, Study Director — University of Sao Paulo General Hospital
Locations (1):
- Hospital das Clinicas of the Medicine College of the University of São Paulo, São Paulo, São Paulo, Brazil